CLINICAL TRIAL: NCT00847093
Title: Post-Operative Pain Control in Children and Infants Undergoing Penoplasty: A Randomized Control Trial of a Local Anesthetic Cream Placebo.
Brief Title: LMX-4 for Postoperative Pain Management in Infants and Children Undergoing Penoplasty Surgery
Acronym: LMX-4
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ferndale Laboratories, Inc. (Industry)
Responsible Party: Santhanam Suresh, MD, Children's Memorial Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: LMX-944700
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2009-02

CONDITIONS: Post-Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cream (Experimental): Experimental group receiving either medicated topical cream or placebo cream
  Interventions: Drug: LMX4; Drug: LMX4 Placebo

INTERVENTIONS:
Drug: LMX4 — One inch every six hours
Drug: LMX4 Placebo — One inch every six hours
  Other Names: Placebo cream

SUMMARY:
After surgery on his penis, your child will probably have some pain. The investigators will give you a prescription for acetaminophen (Tylenol) with codeine, given by mouth (orally), for pain. In this study, the investigators want to see if a local anesthetic cream applied to the base of the shaft of the penis can reduce the need for oral medicine .

DETAILED DESCRIPTION:
Your child will receive a general anesthetic for the surgery. After your child is asleep, he will receive a local anesthetic injection in the area of the tailbone (normal procedure for this surgery). At the end of the operation your child will go to the recovery room. At the time of discharge from the hospital, we will be give you the prescription for acetaminophen with codeine (standard medication given for children undergoing surgery on the penis), and a tube of cream. The tube will contain either a local anesthetic cream (LMX-4)® or a cream with no active medicine (a placebo). We want you to apply the cream to the base of your son's penis every six hours. Which kind of tube you get will be picked randomly (similar to drawing numbers out of a hat) by a computer. Thirty minutes after applying the study cream, or sooner if needed, if you think your child needs pain medication, you may give the oral pain medicine (Tylenol with codeine as prescribed on the bottle). You may continue to apply the cream and give oral medicine every six hours as long as you think your child needs pain medicine for a maximum of 7 days. The cream can also be re-applied when changing diapers to facilitate the continued use of the cream even if it is sooner than the suggested 6 hours.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 3 months to less than 3 years of age (at least 3 months old but not yet reached his 3rd birthday at the time of enrollment).
* Subject has presented with a clinical diagnosis of buried penis
* With the exception of the disease being studied, subject is in good health in the opinion of the investigator.
* Subject and parent(s) or legal guardian(s) must agree to the requirements and restrictions of the study and will appear for all required examinations.
* Subject's parent or legal guardian must sign a written, IRB-approved informed consent prior to admission into the study, and must be able to understand that consent form.

Exclusion Criteria:

* Subject has a known hypersensitivity to any component of the study medication.
* Subject has history or evidence of other conditions that would interfere with evaluation of the study medication.
* Subject has been treated with another investigational device or drug within 30 days prior to study enrollment, or is participating in a clinical trial at the time of enrollment or intends to participate in a clinical trial concurrent with this study.

Ages: 3 Months to 3 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Reducing by 50% the need for rescue analgesia between the LMX4 cream or placebo cream group | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Santhanam Suresh, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Children's Memorial Hospital, Chicago, Illinois, United States